CLINICAL TRIAL: NCT02856256
Title: Study of the Choroidal Thickness Variations After Ingestion of RedBull® Energy Drink
Acronym: REDCHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MMT_2015_2
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Choroid
Keywords: Energy drink; Choroid

ARMS (1):
- RedBull® energy drink (Experimental)
  Interventions: Dietary Supplement: RedBull® energy drink

INTERVENTIONS:
Dietary Supplement: RedBull® energy drink — Subjects consume 25 mL of RedBull® energy drink

SUMMARY:
The choroid is a richly vascularized conjunctive tissue, providing the nutritive elements to the pigmentary epithelium and the photoreceptors of the retina. It drains 80% of the eye's blood. The choroidal thickness fluctuates according to the state of fullness of its constitutive vessels. The choroid and the neuroretina (separate by the pigmentary epithelium) are intimately linked and are subject to modifications during the ingestion of caffeine and taurine combined. Several authors have shown a significant decrease of the choroidal thickness lasting at least 4 hours after the ingestion of a small coffee. This decrease may be caused by caffeine's vasoconstrictor effect. Taurine is the most abundant amino acid in the retina. Recent studies have shown the importance of this amino acid in the physiology of both, retinal pigmentary epithelium and retinal ganglion cells.

RedBull® is an energizing drink, where one single 25 cl can contains 80 mg of caffeine (the equivalent of a coffee mug) and 1 g of taurine.

This pilot trial aims to study the variations of the choroidal thickness and to describe possible modifications within the pigmentary epithelium, due to the ingestion of caffeine and taurine. The results of this study will act as a reference for an ulterior trial aiming specific choroidal pathologies of young patients, such as the central serous chorioretinitis.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-45 years old
* subject under no medical treatment who can alter choroidal depth (sildenafil, diuretics, steroids, etc)
* Non smoker
* subject who has not ingested any caffeine within the 12 hours prior to the trial's inclusion
* subject well informed of the trial and having signed consent

Exclusion Criteria:

* subject with retinal and/or choroidal abnormalities
* Diabetic subject
* Hypermetropia > +3 diopters and myopia < -3 diopters
* History of intra-ocular surgery or laser
* subject with a history of retinal pathologies
* Subject not affiliated to French social security
* Subject under juridical protection
* Pregnant woman

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2017-05-29 (Actual); Study Completion 2017-05-29 (Actual)

PRIMARY OUTCOMES:
Intra-patient variation of the choroidal thickness | up to 4 hours
  Measure of choroidal thickness by Optical Coherence Tomography (OCT), 5 minutes before ingesting 25cl RedBull® then 5 minutes, 30 minutes, 1 hour, 2 hours and 4 hours after ingestion of RedBull®.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France

REFERENCES:
- [Derived] Arej N, Azar G, Salviat F, Alonso AS, Zuber K, Metten MA, Salomon L, Vasseur V, Mauget-Faysse M. Study of choroidal thickness variations after ingestion of a taurine and caffeine-containing energy drink. Clin Nutr ESPEN. 2021 Jun;43:245-249. doi: 10.1016/j.clnesp.2021.04.007. Epub 2021 Apr 17. PMID 34024522